CLINICAL TRIAL: NCT01262586
Title: Pilot Study to Assess the Difference in Glycemic Profiles Between Vildagliptin and Glimepiride Using Continuous Glucose Monitoring Device
Brief Title: Vildagliptin Glycemic Profiles Assessment Using a Continuous Glucose Monitoring Device.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237A23151; 2010-021236-34 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Type II Diabetes Mellitus
Keywords: Type II Diabetes Mellitus; Vildagliptin; Glimepiride; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; glimepiride

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: Vildagliptin
- Glimepiride (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Vildagliptin
  Arms: Vildagliptin
Drug: Glimepiride
  Arms: Glimepiride

SUMMARY:
This study will use Continuous Glucose Monitoring to assess differences in glycemic profiles between vildagliptin and glimepiride.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients on stable metformin
* 18-70 years old
* Willing to perform at least 4 capillary blood glucose tests per day

Exclusion Criteria:

* Type 2 diabetes patients on any other antidiabetic treatment
* Patients listed in other trials
* Patients with significant diabetic organ disease or complications.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in Glycemic profiles between vildagliptin and glimepiride | Baseline and treatment Day 5, 24hr continuous glucose measurements

SECONDARY OUTCOMES:
Glucose Fluctuation before and during treatment | Baseline and treatment Day 5, 24hr continuous measurements

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Mainz, Germany

REFERENCES:
- [Result] He YL, Foteinos G, Neelakantham S, Mattapalli D, Kulmatycki K, Forst T, Taylor A. Differential effects of vildagliptin and glimepiride on glucose fluctuations in patients with type 2 diabetes mellitus assessed using continuous glucose monitoring. Diabetes Obes Metab. 2013 Dec;15(12):1111-9. doi: 10.1111/dom.12146. Epub 2013 Jul 14. PMID 23782529